CLINICAL TRIAL: NCT01807533
Title: A Family-Centered Intervention Program for Preterm Infants: Effects and Their Biosocial Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201103075RB
Record Dates: First submitted 2013-01-29; First posted 2013-03-08 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2017-03

CONDITIONS: Premature Birth
Keywords: Environment; Gene; Intervention; Neurodevelopment; Pathways; Preterm infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-centered intervention program (Experimental): FCIP: family members were encouraged to present in all intervention sessions included 5 in-hospital intervention, 7 after-discharge interventions (0, 1, 2, 4, 6, 9, and 12 months of corrected age), and neonatal follow-up at 0, 1, 6, 12, 18, and 24 months of corrected age.
  Interventions: Behavioral: Family-centered intervention program
- Usual care intervention program (Other): UCP: family members were invited to present at least one session of the 5 in-hospital intervention session. Parents and infants in the UCP group received 7 after-discharge phone calls (0, 1, 2, 4, 6, 9, and 12 months of corrected age) and neonatal follow-up at 0, 1, 6, 12, 18, and 24 months of corrected age.
  Interventions: Behavioral: Usual care intervention program

INTERVENTIONS:
Behavioral: Family-centered intervention program — This program was in-hospital intervention, after-discharge intervention, and neonatal follow-up. Five sessions of in-hospital intervention emphasized in the parental involvements with modulation of the NICU, a teaching of child developmental skills, feeding support, massage, interactional activities, child developmental skills, parent support and education, and transition home preparation. The 7-session after-discharge intervention consisted of 4 clinic visits and 3 home visits with specific care in modulation of home environment, teaching of child developmental skills, feeding support, teaching of interactional activities, and parent support and education
  Other Names: FCIP
  Arms: Family-centered intervention program
Behavioral: Usual care intervention program — This program was in-hospital intervention, after-discharge consultation, and neonatal follow-up. Five sessions of in-hospital intervention emphasized in the parental involvements with modulation of the NICU, a teaching of child developmental skills, feeding support, massage, interactional activities, child developmental skills, parent support and education, and transition home preparation. The after-discharge service was provided 7-phone calls for the general health consultation.
  Other Names: UCP
  Arms: Usual care intervention program

SUMMARY:
Four hypotheses will be tested in this study:

1. The intervention group performs better in child, parent and transactions outcomes than the control group throughout the follow-up period.
2. The intervention group shows greater changes in early neurophysiological brain functions and transactions within the family that lead to better neurodevelopmental outcomes than the control group.
3. Certain polymorphisms of the dopamine-related genes are associated with the neurodevelopmental outcomes in VLBW preterm infants.
4. Very low birth weight preterm infants carrying more genetic plasticity in the dopamine-related genes may benefit more from the interventions than those carrying less genetic plasticity.

DETAILED DESCRIPTION:
A total of 275 VLBW preterm infants (269 participants and 6 pilots) were recruited at three medical centers in northern and southern Taiwan and were randomly assigned to the FCIP or UCP group. Outcome assessments included primary (neurobehavioral development) and secondary measures (neurophysiological performance, parents' stress and transactions within the family). The neurophysiological and transactions data were examined for whether they mediate intervention effects on child development. In addition, these infants 219 VLBW preterm infants and 118 term infants in our prior intervention studies were collected buccal cells for assessment of the polymorphisms of dopamine-related genes, which are involved in the neurotransmission of cognitive, sensorimotor and behavioral-emotional systems and postulated to be associated with several developmental and psychiatric illnesses. The polymorphisms of dopamine-related genes were examined for potential moderating influence on the effects of the intervention for child development.

ELIGIBILITY:
Inclusion Criteria:

* birth body weight < 1500 grams
* gestational age < 37 weeks
* parents of Taiwan nationality, married or together at delivery, and northern family residing in greater Taipei and southern family residing in greater Tainan, Kaohsiung, or Chiayi

Exclusion Criteria:

* severe neonatal and perinatal diseases (e.g., seizures, hydrocephalus, meningitis, grade III-IV IVH and grade II NEC)
* congenital or chromosome abnormality
* mother < 18 years, with mental retardation or history of maternal substance abuse at any time (smoking, alcohol, and drug)

Terminated Criteria:

* diagnosis of brain injury (e.g., PVL, stage IV ROP or greater)
* severe cardiopulmonary disease requiring invasive or non-invasive ventilator use at hospital discharge
* hospital discharge beyond 44 weeks' post-menstrual age.

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2012-05-22 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Child: neurodevelopment functions (cognition, language and motor) | 24 months of corrected age
  Bayley Scales of Infant and Toddler Development - 2nd and 3rd edition

SECONDARY OUTCOMES:
Change of neurodevelopment functions (motor) from baseline | 0 months of corrected age
  The Neonatal Neurobehavioral Examination-Chinese Version (NNE-C) 2. World Health Organization Quality of Life- Brief Taiwan version
Child: neurodevelopment functions (behavior) | 24 months of corrected age
  Child behavior checklist version 1.5-5 Y 2. World Health Organization Quality of Life- Brief Taiwan version
Change of neurodevelopment functions (cognition, language and motor) from baseline | 6,12, and 24 months
  Bayley Scales of Infant and Toddler Development - 3rd edition 2. World Health Organization Quality of Life- Brief Taiwan version
Parental functions and change from baseline (pressure) | 0, 6, 12, 18, and 24 months of corrected age
  Parenting Stress Index 2. World Health Organization Quality of Life- Brief Taiwan version
Parental functions and change from baseline (Quality of Life) | 0, 6, 12, 18, and 24 months of corrected age
  World Health Organization Quality of Life- Brief Taiwan version
Transactional functions and change from baseline | 6, 12, and 18 months of corrected age
  Mother-infant interaction in free play at 6, 12, and 18 months of corrected age
Transactional functions and change from baseline | 6 and 12 months of corrected age
  Wakeful Position Questionnaire at 6 and 12 months of corrected age
Transactions function: affordance | 18 months of corrected age
  1. Affordances in the Home Environment Motor Development- Chinese version
Child: Medical data | Birth to 24 months of corrected age
  Chart review
Child: growth data and change from baseline | 0, 1, 4, 6, 12, 18, and 24 months of corrected age
  Chart review and measurement
Child: neurophysiological functions and change from baseline | 1 and 4 months of corrected age
  Electroencephalogram/event-related potential
Child: genotyping and gene expression | 0 month of corrected age
  Buccal cell collection
Parental adherence to Intervention | 32-36 weeks (5 sessions), 0, 1, 2, 4, 6, 9, and 12 months
  Only assessed in FCIP group
  1. Parental motivation
  2. Goal attainment
  3. Home activity records

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Fang Jeng, Professor, Principal Investigator — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (3):
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li SJ, Tsao PN, Tu YK, Hsieh WS, Yao NJ, Wu YT, Jeng SF. Cognitive and motor development in preterm children from 6 to 36 months of age: Trajectories, risk factors and predictability. Early Hum Dev. 2022 Sep;172:105634. doi: 10.1016/j.earlhumdev.2022.105634. Epub 2022 Jul 28. PMID 35921693
- [Derived] Yu YT, Huang WC, Hsieh WS, Chang JH, Lin CH, Hsieh S, Lu L, Yao NJ, Fan PC, Lee CL, Tu YK, Jeng SF. Family-Centered Care Enhanced Neonatal Neurophysiological Function in Preterm Infants: Randomized Controlled Trial. Phys Ther. 2019 Dec 16;99(12):1690-1702. doi: 10.1093/ptj/pzz120. PMID 31504897